CLINICAL TRIAL: NCT02405767
Title: Characterisation by Electric Impedance Measurements of the Different Wound Healing Phases of Diabetic Foot Ulcers
Brief Title: BioimPEDance of Diabetic Foot Ulcers
Acronym: BIPPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Grenoble University Hospital.; 2015-A00070-49 (Other: ID RCB)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foot ulcer impedance (Experimental): Diabetic patients with a diabetic foot ulcer
  Interventions: Other: Foot ulcer impedance

INTERVENTIONS:
Other: Foot ulcer impedance — lmpedence measured using ECG electrodes placed at the periphery of the wound (when the wound dressing is changed as part of standard care).

SUMMARY:
The BIPPED study seeks to determine whether wound healing, in particular diabetic foot ulcers, can be monitored using electrical bioimpedance analysis (BIA). BIA measures the resistance of biological tissue to the passage of a very small electric current applied with electrodes. Different types of tissue, due to cell structure, hydration and vascularization, have specific electrical characteristics. The BIPPED study aims to provide experimental data for the development of a BIA sensor for monitoring of wound healing in chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patient (Type 1 or 2) with diabetic foot ulcer or lower limb ulcer
* written informed consent signed
* insured by the French national health insurance scheme

Exclusion Criteria:

* wound in the similar position on the other limb
* people under legal protection
* unilateral limb oedema
* contra-indication to impedancemetry : pregnancy, patient with a pacemaker, neurostimulator or any other implanted electrical device, metallic prostheses
* patients participating to other protocols involving foot ulcers measurement, if it interfers with the current protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09-02 (Actual); Study Completion 2016-09-02 (Actual)

PRIMARY OUTCOMES:
Change in impedance | 3 months
  Correlation between electrical impedance of the wound measured with ECG electrodes placed at the periphery of the wound and changes in the size of the wound and the clinically observed stage of healing.

SECONDARY OUTCOMES:
Impedance of different wound tissues | 3 months
  Characteristic impedance of different types of wound tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France

REFERENCES:
- [Background] Lukaski HC, Moore M. Bioelectrical impedance assessment of wound healing. J Diabetes Sci Technol. 2012 Jan 1;6(1):209-12. doi: 10.1177/193229681200600126. PMID 22401341